CLINICAL TRIAL: NCT03774043
Title: Timing and Dosage Parameters of Acute Intermittent Hypoxia in Individuals With Spinal Cord Injury.
Brief Title: Timing and Dosage of Acute Intermittent Hypoxia in Persons With SCI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Milap Sandhu, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00202027
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Single session of Acute Intermittent Hypoxia (AIH) (Experimental)
  Interventions: Other: Acute Intermittent Hypoxia
- Single session of Sham Acute Intermittent Hypoxia (Sham AIH) (Placebo Comparator)
  Interventions: Other: Sham Acute Intermittent Hypoxia
- Two successive sessions of AIH (Experimental)
  Interventions: Other: Acute Intermittent Hypoxia
- Two successive sessions of Sham AIH (Placebo Comparator)
  Interventions: Other: Sham Acute Intermittent Hypoxia

INTERVENTIONS:
Other: Acute Intermittent Hypoxia — Patients will breath 9%-11% oxigen for 1.5 minutes interspersed with 1.5 minutes of 21% oxigen (normoxia), 15 times for a total of 45 minutes.
  Arms: Single session of Acute Intermittent Hypoxia (AIH); Two successive sessions of AIH
Other: Sham Acute Intermittent Hypoxia — Patients will breath 21% oxigen for 1.5 minutes interspersed with 1.5 minutes of room air, 15 times for a total of 45 minutes.
  Arms: Single session of Sham Acute Intermittent Hypoxia (Sham AIH); Two successive sessions of Sham AIH

SUMMARY:
This study will utilize short duration and mild levels of reduced oxygen (hypoxia) to induce spinal plasticity while evaluating the appropriate timing schedule for this intervention, as well as, the effects of superimposing sessions of a therapy, in individuals with chronic incomplete SCI. Our aim is to establish the time-course of outcome improvement and decay following a single session or multiple sessions of AIH therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Spinal cord lesion at level of C3 to T1
2. Individuals with a history of incomplete spinal cord injury, classified as ASIA C or D
3. Individuals must be at least 6 months status post injury
4. Individuals must be between the ages of 18-70 years inclusive, male or female
5. Spinal cord injury must be secondary to a non-progressive etiology
6. Individuals must be medically stable.
7. Able to comply with protocol/study requirements
8. Not currently (>2 weeks) taking any medications for spasticity management.

Exclusion Criteria:

1. Recent change in the use of narcotic, anti-inflammatory or pain medication
2. Unstable medical conditions or any other clinical observation that may affect the candidate's performance, health, safety or the ability to participate in the study, as determined by the treating therapist
3. History of sleep apnea
4. Active participation in another movement research study or therapy program
5. Anti-spasticity drug injection less than 3 months, prior to beginning treatment
6. Musculoskeletal pain that interferes with participation in study
7. Women who are currently, may be or planning on becoming pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-03 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in grip strength | Baseline, immediately following intervention, and every 30 minutes for 5 hours
  A dynamometer measures maximum gross grasp (kglb) averaged over three attempts with each hand. The minimum possible value of zero kg lb will be assigned when the participant cannot actively flex the fingers or grasp the dynamometer. Standard position includes the participant in a supported sitting position, with shoulder in adducted and in neutral rotation and the elbow flexed at 90 degrees. The forearm should be in neutral rotation. The arm should not be supported by an arm rest or research personnel.
Pinch Strength | Baseline, immediately following intervention, and every 30 minutes for 5 hours
  A pinch gauge measures maximum pinch force (kglb) averaged over three attempts with each hand. The minimum possible value of zero kg will be assigned when the participant cannot actively squeeze the pinch meter between the thumb and index finger. Standard position includes the participant in a supported sitting position, with shoulder in adducted and in neutral rotation and the elbow flexed at 90 degrees. The gauge will be placed between the thumb and lateral surface of the index finger (lateral pinch).
9 Hole Peg Test | Baseline, immediately following intervention, and every 30 minutes for 5 hours
  A measure of finger dexterity involving the placement of pegs from a container to holes on a board, and subsequent removal, as quickly as possible. The total number of seconds until task completion is recorded, as measured by when the participant touches the first peg to when the last peg is placed back into the container.
Box and Blocks test | Baseline, immediately following intervention, and every 30 minutes for 5 hours
  A measure of manual dexterity that requires repeatedly moving 1-inch blocks from one side of a box to another in 60 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States